ClinicalTrials.gov ID: NCT03483961

Document: PXVX-CV-317-001 IRB-Approved Site Informed Consent Form

Informed Consent Form (ICF) Version: v3.0

Informed Consent Form (ICF) Version Date: 06-June-2019

Informed Consent Form (ICF) IRB Approval Date: 06-June-2019